CLINICAL TRIAL: NCT04779931
Title: The Usability and Feasibility of Social Convoy Palliative Care (Convoy-Pal) Mobile Health for Older Adults
Brief Title: Social Convoy Palliative Care (Convoy-Pal) Mobile Health for Older Adults
Acronym: ConvoyPal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18-0973; K76AG059934 (NIH)
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Chronic Conditions, Multiple
MeSH Terms: conditions — Multiple Chronic Conditions

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convoy-Pal Intervention (Experimental): Intervention participants will be sent Convoy-Pal equipment and materials. The equipment can simply be removed from the box, plugged in, and turned on to start. Research staff will provide technical support as needed during the trial. Convoy-Pal is 12-week intervention that uses the Routinify platform to deliver self-management tools and palliative care resources in the participants' home. The platform includes a tablet, charging stand, and smart watch, with additional options for mobile phone access and a website portal.
  Interventions: Behavioral: Convoy-Pal
- Waitlist Control (Active Comparator): Participants will complete baseline assessments and will be recontacted at 11 weeks to complete follow up assessments at week 12. Participants will receive a $25 gift card for each assessment ($50 total). If they would like to try the intervention at that time, we will send them Convoy-Pal equipment and materials. They will then have 12 weeks to use the tool.
  Interventions: Behavioral: Convoy-Pal

INTERVENTIONS:
Behavioral: Convoy-Pal — 12 week mobile self-management intervention with palliative care resources.

SUMMARY:
The aim of this study is to test the feasibility and usability of the Convoy-Pal mobile intervention among older adults. The study is a pilot waitlist control RCT with 40 patients and their convoys randomized to one of two arms: Convoy-Pal intervention or waitlist control. Feasibility will be assessed by recruitment, attrition, and data collection on measures of quality of life and social support. Usability will be captured by self-report usability scales and actual back end utilization data.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* self-report diagnosis of heart failure (HF)
* have multiple chronic conditions (MCC) based on the Disease Burden/Morbidity Assessment by Self-Report (Individuals will be eligible if they self-report the number of diagnosis > 2 and a disease burden score >2 indicating the presence of at least two chronic conditions that limit activities of daily of living)
* community dwelling in the United States
* English speaking

Exclusion Criteria:

* Self-reported diagnosis of Alzheimer's disease or dementia
* Self-reported diagnosis of a severe mental health problem (e.g. schizophrenia, bipolar affective disorder or other psychotic illness)
* Participation in community-based palliative care in the last 12 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
User Mobile Application Rating Scale | 12 weeks
  Usability; 20 items; Range 0-25, Higher score indicates better usability

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer D Portz, PhD, MSW, Principal Investigator — University of Colorado Denver | Anschutz
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] DeGroot L, Gillette R, Villalobos JP, Harger G, Doyle DT, Bull S, Bekelman DB, Boxer R, Kutner JS, Portz JD. Feasibility of a digital palliative care intervention (Convoy-Pal) for older adults with heart failure and multiple chronic conditions and their caregivers: a waitlist randomized control trial. BMC Palliat Care. 2024 Oct 1;23(1):234. doi: 10.1186/s12904-024-01561-w. PMID 39354453